CLINICAL TRIAL: NCT06652139
Title: A Single-center, Randomized Controlled Clinical Study of Selinexor Combined With BEAM as a Preconditioning Regimen for ASCT in Relapsed and Refractory Diffuse Large B-cell Lymphoma With MYC Positive
Brief Title: Selinexor Combined With BEAM for ASCT in R/R DLBCL With MYC Positive
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SINE+BEAM
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B cell lymphoma; Autologous stem cell transplantation; Selinexor; BEAM
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — BEAM regimen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selinexor combined with BEAM pretreatment regimen (Experimental): Patients in this arm will receive selinexor combined with BEAM (carmustine, etoposide, cytarabine and melphalan) as pretreatment regimen of ASCT.
  Interventions: Drug: selinexor combined with BEAM regimen
- BEAM pretreatment regimen (Active Comparator): Patients in this arm will receive BEAM (carmustine, etoposide, cytarabine and melphalan) as pretreatment regimen of ASCT.
  Interventions: Drug: BEAM regimen

INTERVENTIONS:
Drug: selinexor combined with BEAM regimen — Selinexor: 60mg po D-10, D-7 and D-4 Carmustine: 300mg/m2 ivgtt D-8 Etoposide: 100mg/m2/d ivgtt q12h D-7-D-4 Cytarabine: 200mg/m2/d ivgtt q12h D-7-D-4 Melphalan: 140mg/m2 ivgtt D-3-D2
  Other Names: SINE+BEAM
  Arms: selinexor combined with BEAM pretreatment regimen
Drug: BEAM regimen — Carmustine: 300mg/m2 ivgtt D-8 Etoposide: 100mg/m2/d ivgtt q12h D-7-D-4 Cytarabine: 200mg/m2/d ivgtt q12h D-7-D-4 Melphalan: 140mg/m2 ivgtt D-3-D2
  Other Names: BEAM
  Arms: BEAM pretreatment regimen

SUMMARY:
To evaluate the efficacy and safety of selinexor combined with BEAM pretreatment regimen in ASCT of recurrent and refractory DLBCL patients with immunohistochemical positive for MYC

DETAILED DESCRIPTION:
This trial included 82 patients, who were randomly divided into pre-treatment with selinexor combined with BEAM regimen (experimental group) or BEAM regimen (control group) according to 1:1, and then underwent ASCT therapy. The trial included a screening period, a treatment period (2 weeks before and after transplantation), and a follow-up period (2 years after autologous transplantation). At 3, 6, 9 and 18 months after ASCT, blood routine, blood biochemistry, B-ultrasound of liver, bile, pancreas, spleen and lymph node, and whole body enhanced CT were performed. At 1 and 2 years after ASCT, blood routine, blood biochemistry, and whole body PET-CT evaluation were performed until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. According to world Health Organization (WHO) classification of disease, diffuse large B-cell lymphoma was confirmed by histology, CR or PR after second-line and above treatment;
2. The subjects tested positive for MYC in primary or pre-transplant lymphoma lesions;
3. 18≤ age ≤65 years old, male or female;
4. ECOG score 0-2;
5. No serious organic lesions in the main organs, meeting the requirements of the following laboratory examination indicators (conducted within 7 days before treatment) :

   1. White blood cell count ≥3.0×109/L, absolute neutrophil count ≥1.5×109/L, Hemoglobin ≥90g/L, platelet ≥75×109/L;
   2. Total bilirubin ≤1.5× upper normal value (ULN);
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× ULN; Bilirubin ≤1.5× ULN
   4. Creatinine clearance was 44-133 mmol/L;
6. No cardiac dysfunction;
7. Life expectancy over 3 months;
8. The subject or his/her legal representative must provide written informed consent prior to conducting a special study examination or procedure.

Exclusion Criteria:

1. Previously received autologous hematopoietic stem cell transplantation;
2. Suffering from serious complications or severe infection;
3. Previous treatment with selinexor;
4. Central nervous system lymphoma was excluded;
5. A history of other malignant tumors within 5 years, excluding early tumors treated for curative purposes;
6. Patients with uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc.;
7. HBsAg, HCV or HIV positive. Positive HBV and HCV serology is allowed, but DNA/RNA testing must be negative;
8. Left ventricular ejection fraction ≦ 50%;
9. Laboratory test value during screening;

   ① Neutrophils <1.5×109/L; Platelet <75×109/L;

   ② Bilirubin was 1.5 times higher than the normal upper limit, transaminase was 2.5 times higher than the normal upper limit;

   ③ The creatinine level is higher than 1.5 times the upper limit of normal value;
10. Other concurrent and uncontrolled medical conditions considered by the investigator would affect the patient's participation in the study;
11. Psychiatric patients or other patients known or suspected to be unable to fully comply with the study protocol;
12. Pregnant or lactating women;
13. The researcher judged that the patients were not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of ASCT until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from an cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of ASCT to the date of death from any cause.
Complete remission rate | 3 months after the transplantation
  Percentage of participants with complete response was determined on 2014 Lugano criteria.
The time of hematopoietic reconstruction | 2 months after the transplantation
  The first day of neutrophils ≥0.5×109/L for 3 consecutive days was the time of successful implantation of granulocytes. Platelet ≥20.0×109/L for 7 consecutive days and the first day after platelet infusion was considered as the successful time of megakaryocytes implantation.
Transplantation-related adverse reactions | Baseline up to data cut-off (up to approximately 4 years)
  Transplantation-related adverse reactions are any untoward medical occurrence in a participant which is related to ASCT.

IPD SHARING:
Plan to Share IPD: No